CLINICAL TRIAL: NCT04502810
Title: A Feasibility and Acceptability Study of High-level Laser for Women With Provoked Vestibulodynia
Brief Title: High-level Laser for Provoked Vestibulodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Exogenia (Unknown)
Responsible Party: Principal Investigator, Mélanie Morin, Researcher and Associate Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #2020-3535
Record Dates: First submitted 2020-07-27; First posted 2020-08-06 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Vulvodynia
Keywords: Laser; Provoked vestibulodynia; Pain; Sexual dysfunctions
MeSH Terms: conditions — Vulvodynia; Pain

STUDY DESIGN:
Intervention Model Description: Baseline evaluation - Randomization to real laser or sham laser (12 sessions in 6 consecutive weeks) - Post-treatment evaluation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-level laser therapy (Experimental): Real high-level laser therapy laser 12 biweekly sessions (6 consecutive weeks of biweekly treatments)
  Interventions: Radiation: High-level laser therapy
- Sham High-level laser therapy (Sham Comparator): Sham high-level laser therapy laser 12 biweekly sessions (6 consecutive weeks of biweekly treatments)
  Interventions: Radiation: High-level laser therapy

INTERVENTIONS:
Radiation: High-level laser therapy — Nd:Yag 1064 nm pulsed high-level Laser will be applied to the vulvar area.
  Other Names: Nd:Yag laser

SUMMARY:
This is a randomized feasibility and acceptability study investigating the effects of laser treatment in women suffering from provoked vestibulodynia compared to a sham-laser treatment. Participants will be randomized into the laser group or sham-laser group. The laser group will receive 12 sessions of real high-level laser therapy (HILT) (30-minutes biweekly for 6 consecutive weeks). The sham-laser group will receive 12 sessions (30-minutes biweekly for 6 consecutive weeks) of laser therapy using a deactivated probe. Outcomes measures will be assessed at baseline and at post-treatment and will include: feasibility and acceptability variables, pain, sexual function, sexual distress, psychological variables and perceived improvement after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe pain (≥5/10) during sexual intercourse for at least 3 months
* Moderate to severe pain (≥5/10) in at least 90% of sexual intercourses or attempted sexual intercourse for at least 3 months
* Provoked vestibulodynia lasting at least 3 months prior to the study and diagnosed by a standardised gynaecologic exam

Exclusion Criteria:

* Other causes of vulvo-vaginal pain (e.g. spontaneous vulvovaginal pain not related to sexual intercourse/contact, dermatological condition, herpes, vulvo-vaginal atrophy)
* Post-menopausal state
* Actual or past pregnancy in the last year
* Urogynecological condition (e.g. pelvic organs prolapse ≥3, urinary/vaginal infection active or in the last 3 months)
* Anterior vulvar, vaginal or pelvic surgery (e.g. vestibulectomy, corrective pelvic organs prolapses surgery)
* Prior use of laser treatments for vulvar pain
* Expected changes of medication that could influence pain perception (e.g. analgesic, antidepressant)
* Other medical conditions that could interfere with the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Adherence rate | 2-week post-treatment evaluation
  To determine acceptability by assessing adherence to treatment sessions
Level of satisfaction with the treatment | 2-week post-treatment evaluation
  To determine acceptability by measuring the participants' satisfaction with the treatment on a numeric rating scale ranging from 0 (completely dissatisfied) to 10 (completely satisfied)
Willingness to recommend the treatment | 2-week post-treatment evaluation
  To determine acceptability by assessing whether the participant would recommend the treatment.
Rate of adverse events | 2-week post-treatment evaluation
  To document any adverse events.
Blinding effectiveness | 2-week post-treatment evaluation
  To assess the feasibility of maintaining blinding to group allocation for the therapists, assessors and therapists. Evaluated by asking the question: ''What treatment do you think you have received / given? ''
Recruitment rate | Baseline to 2-week post-treatment evaluation
  To assess the recruitment rate including the barriers and reasons for refusing to participate as well as the reasons for exclusion
Completion and dropout rates | 2-week post-treatment evaluation
  To evaluate completion and dropout rates based on the completion of the post-treatment evaluation.
Completeness of data | Baseline to 2-week post-treatment evaluation
  To examine the percentage of completed outcome measures.

SECONDARY OUTCOMES:
Change in pain intensity during intercourse | Baseline to 2-week post-treatment evaluation
  To explore changes in pain intensity during intercourse (Numerical Rating Scale, ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain ever)
Change in sexual function | Baseline to 2-week post-treatment evaluation
  To explore changes in sexual function (Female Sexual Function Index). Minimum value: 2, Maximum value: 36 and lower scores mean worst outcome (low sexual function).
Change in sexual distress | Baseline to 2-week post-treatment evaluation
  To explore changes in sexual distress (Female Sexual Distress Scale ). Minimum value: 0, Maximum value: 52, higher scores mean worst outcome (higher sexually related distress).
Change in pain quality | Baseline to 2-week post-treatment evaluation
  To explore changes on the sensory, affective and evaluative components of pain (McGill-Melzack Questionnaire). Minimum value: 0, Maximum value: 78, higher scores mean worst outcome (higher pain).
Patient's global impression of change | Baseline to 2-week post-treatment evaluation
  To examine patient self-reported improvement (Patient's Global Impression of Change ranging from "very much worse" to "very much improved" on a 7-point scale.
Change in fear of pain | Baseline to 2-week post-treatment evaluation
  To explore changes in fear of pain (Pain Anxiety Symptoms Scale (PASS-20)). Minimum value: 0, Maximum value: 100, higher scores mean worst outcome (higher fear of pain).
Change in pain catastrophization | Baseline to 2-week post-treatment evaluation
  To explore changes in pain catastrophization (Pain Catastrophizing Scale (PCS)). Minimum value: 0, Maximum value: 52, higher scores mean worse outcome (higher pain catastrophization)
Change in vulvar pain sensitivity | Baseline to 2-week post-treatment evaluation
  To explore changes in vulvar pain sensitivity (algometer)
Change in vulvar blood circulation | Baseline to 2-week post-treatment evaluation
  To explore changes in vulvar blood circulation using the laser speckle. Vulvar vestibule blood perfusion is expressed in arbitrary perfusion units (APUs).

CONTACTS AND LOCATIONS:
Overall Officials: Mélanie Morin, PT, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier Universitaire de Sherbroke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No